CLINICAL TRIAL: NCT00346060
Title: Safety Study in Retinal Transplantation for Dry Age Related Macular Degeneration.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radtke, Norman D., M.D. (Individual)
Collaborators: Foundation Fighting Blindness (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 20050380
Record Dates: First submitted 2006-06-28; First posted 2006-06-29 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Dry Age Related Macular Degeneration.
Keywords: Dry age related macular degeneration.; Retinal Transplant; Fetal Tissue; Early treatment diabetic retinopathy study; 20/200 or worse.

INTERVENTIONS:
Device: Retinal transplantation instrument
Device: Fetal tissue.

SUMMARY:
The long-term goal is to show that retinal transplantation can help to prevent blindness and to restore eyesight in patients with dry age related macular degeneration.

DETAILED DESCRIPTION:
The aim of this clinical trial is to test the safety of transplanting human fetal neural retinal tissue and retinal pigment epithelium into the eyes of human patients with age-related macular degeneration. Vision in the eye to be operated on will be the poorer vision of both eyes and must be 20/200 or worse. "Retinal tissue", the layers in the back of the eye, consists of neural retina and retinal pigment epithelium. "Neural retina" is the nerve cell layer that processes light into vision. The "photoreceptor cells" in the neural retina detect the light and transform it into electrical signals, which are then transferred to the brain by other retinal cells. "Retinal pigment epithelium" (RPE) is the layer behind the neural retina which helps both to nourish the cells of the neural retina and also to get rid of waste products. The fetal tissues used in this study will be derived from dead fetuses in the first 9-16 weeks of pregnancy obtained from elective abortions.

Fetal retinal transplantation is highly experimental. The research will be conducted in accordance with the prohibitions regarding the use of human fetal tissue described in Public Law 103-43, section 498B. There will be no compensation for the donor. The research will be conducted in accordance with any applicable Federal, State and local laws.

First, the technical application of the implantation instrument and its safety in the transplantation will be demonstrated in patients with 20/200 vision in one eye or worse, with functional acuity in the contra lateral eye.

Secondly, the human fetal retinal tissue will be placed in the areas beneath the retina where presently the patient has atrophy of the retinal pigment epithelium and poor retinal function.

ELIGIBILITY:
Inclusion Criteria:

* The subject must have decreased central visual acuity of 20/200 or worse in one eye by ETDRS vision testing for a duration of at least one year in the operated eye and have the diagnosis of age related macular degeneration; vision in the nonoperated eye must be better than the operated eye. Vision in the operated eye cannot be better than 20/200.
* Subject is older than 55 years of age
* Patient is willing to return for follow-up visits
* Patient has signed informed consent for retinal transplantation
* Patient has undergone microperimetry and Goldmann visual field testing.

Exclusion Criteria:

* Patient having a central visual acuity of better than 20/200 in one eye by ETDRS or vision worse than 20/200 in one eye by ETDRS for a duration of less than one year
* Unwilling to sign an informed consent
* Patient under 55 years of age
* Patient having medical problems that are contraindicatory for short-term anesthesia
* Patient unwilling to return for follow-up visits
* The patient has been determined to be pregnant by patient history or by pregnancy testing in women of childbearing potential
* Features of any condition other than age-related macular degeneration in the study eye (such as pathologic myopia or presumed ocular histoplasmosis) associated with choroidal neovascularization
* Any significant ocular disease (other than choroidal neovascularization) that has compromised or could compromise vision in the study eye and confound analysis of the primary outcome.
* Inability to obtain photographs to document choroidal neovascularization, including difficulty with venous access
* History of choroidal neovascularization in the study eye
* Participating in another ophthalmic clinical trial or use of any other investigational new drugs within 12 weeks before the start of study treatment
* Prior photodynamic therapy or Macugen therapy for choroidal neovascularization
* Patient who has a history of uveitis, Coat's disease, diabetic retinopathy, glaucoma, or a cataract that prevents visualization of the posterior pole

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2002-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Snellen
Visual acuity
Microperimetry
Goldmann visual field
Optical coherent tomography
Fluorescein angiography

SECONDARY OUTCOMES:
No rejection of transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Norman D. Radtke, M.D., Principal Investigator — Norman D. Radtke, M.D.
Locations (1):
- Retina Vitreous Resource Center, Louisville, Kentucky, United States

REFERENCES:
- [Result] Radtke ND, Aramant RB, Seiler MJ, Petry HM, Pidwell D. Vision change after sheet transplant of fetal retina with retinal pigment epithelium to a patient with retinitis pigmentosa. Arch Ophthalmol. 2004 Aug;122(8):1159-65. doi: 10.1001/archopht.122.8.1159. PMID 15302656
- [Result] Radtke ND, Seiler MJ, Aramant RB, Petry HM, Pidwell DJ. Transplantation of intact sheets of fetal neural retina with its retinal pigment epithelium in retinitis pigmentosa patients. Am J Ophthalmol. 2002 Apr;133(4):544-50. doi: 10.1016/s0002-9394(02)01322-3. PMID 11931789
- [Result] Radtke ND, Aramant RB, Seiler M, Petry HM. Preliminary report: indications of improved visual function after retinal sheet transplantation in retinitis pigmentosa patients. Am J Ophthalmol. 1999 Sep;128(3):384-7. doi: 10.1016/s0002-9394(99)00250-0. PMID 10511047
- [Result] Radtke ND, Aramant RB, Petry HM, Green PT, Pidwell DJ, Seiler MJ. Vision improvement in retinal degeneration patients by implantation of retina together with retinal pigment epithelium. Am J Ophthalmol. 2008 Aug;146(2):172-182. doi: 10.1016/j.ajo.2008.04.009. Epub 2008 Jun 10. PMID 18547537
- See also: Retina Vitreous Resource Center — http://www.rvrc.com